CLINICAL TRIAL: NCT05304949
Title: Regulatory Post-Marketing Surveillance(PMS) Study for Lucentis®(Ranibizumab) in Patients With Retinopathy of Prematurity
Brief Title: Regulatory PMS Study for Lucentis® in Patients With Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CRFB002HKR01
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; NIS; Post-Marketing Surveillance; Lucentis; Ranibizumab; Korea
MeSH Terms: conditions — Retinopathy of Prematurity | interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Lucentis: Patients prescribed with Lucentis
  Interventions: Other: Lucentis

INTERVENTIONS:
Other: Lucentis — There was no treatment allocation. Patients administered Lucentis by prescription were enrolled.
  Other Names: Ranibizumab

SUMMARY:
This study was an open-labeled, multicenter, single arm, observational post-marketing surveillance study under routine clinical practice with no mandated treatments, visits or assessments.

DETAILED DESCRIPTION:
The investigators collected safety information and evaluated effectiveness in patients who were prescribed with Lucentis® (Ranibizumab) injection in Retinopathy of Prematurity indication after receiving informed consent over a period of 4 weeks.

Subjects who received multiple doses, i.e., 2 or more doses, of Lucentis® injection were defined as subjects with long-term use, and the safety and effectiveness information of up to 12 weeks was collected and analyzed separately.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants with retinopathy of prematurity (ROP)
2. Patients (infants) prescribed with Lucentis® injection according to the product approval information in the Republic of Korea
3. In the case that the legal guardian of the patient (infant) provided a written consent to participate in this study

Exclusion Criteria:

1. In the case that the legal guardian of the patient (infant) does not want participation in this study
2. In the case that it falls under any of the contraindications listed in local prescribing information of Lucentis® injection

   * Patients with hypersensitivity to the active substance or to any of the excipients
   * Patients with an active or suspected ocular or periocular infection.
   * Patients with active intraocular inflammation

Ages: 0 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Korean patients who are prescribed with Lucentis® (Ranibizumab) injection in ROP indication
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2022-06-22 (Actual); Primary Completion 2025-01-11 (Actual); Study Completion 2025-01-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events/adverse drug reactions | Up to 12 weeks
  Incidence of adverse events/adverse drug reactions, serious adverse events/adverse drug reactions, unexpected adverse events/adverse drug reactions, suspected unexpected serious adverse reactions/adverse drug reactions were collected

SECONDARY OUTCOMES:
Proportion of treatment success | Up to 12 weeks
  Proportion of treatment success, defined as regression of proliferative phase and/or complete peripheral retinal vascularization as assessed by the investigator

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- South Korea (3):
  - Novartis Investigative Site, Daegu, Dalseo gu
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CRFB002HKR01 from the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18329